CLINICAL TRIAL: NCT03451110
Title: A 3-Part, Open-label Study to Assess the Pharmacokinetic Drug-Drug Interactions of Lemborexant When Coadministered With an Oral Contraceptive, Famotidine, or Fluconazole in Healthy Subjects
Brief Title: Study to Assess the Pharmacokinetic Drug-Drug Interactions of Lemborexant When Coadministered With an Oral Contraceptive, Famotidine, or Fluconazole in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Collaborators: Purdue Pharma LP (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: E2006-A001-012
Record Dates: First submitted 2018-02-23; First posted 2018-03-01 (Actual); Last update posted 2018-09-06 (Actual); Status verified 2018-02

CONDITIONS: Healthy Subjects
Keywords: Drug-Drug Interactions; Lemborexant; Oral Contraceptive; Famotidine; Fluconazole; Pharmacokinetics; Proton pump inhibitors; CYP3A inhibitors
MeSH Terms: interventions — lemborexant; norethindrone acetate, ethinyl estradiol, ferrous fumarate drug combination; Famotidine; Fluconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1: Lemborexant plus Loestrin (Experimental): Healthy female participants will receive a single oral dose of Loestrin 1.5/30 (containing ethinyl estradiol [EE] 0.030 milligrams [mg] and norethindrone [NE] 1.5 mg) in the evening of Day 1 after a fast of at least 3 hours. After a washout period of at least 4 days, participants will receive 10 mg lemborexant orally for 10 days. Lemborexant will continue to be administered in the evening on Days 15 through 18, followed by a single oral dose of Loestrin on Day 15 when administered with lemborexant after fasting in the evening for at least 3 hours.
  Interventions: Drug: lemborexant; Drug: Loestrin
- Part 2: Lemborexant plus Famotidine (Experimental): Healthy participants will receive a single oral dose of 10 mg lemborexant in the morning of Day 1 after an overnight fast of at least 10 hours. On Day 15, participants will receive a single oral dose of 40 mg famotidine, followed at least 2 hours later by a single dose of 10 mg lemborexant. After a washout period of up to 14 days participants will receive 10 mg lemborexant orally for 10 days.
  Interventions: Drug: lemborexant; Drug: famotidine
- Part 3: Lemborexant plus Fluconazole (Experimental): Healthy participants will receive a single oral dose of 10 mg lemborexant in the morning of Day 1 after an overnight fast of at least 10 hours. After a washout interval of approximately 10 days, on Day 11, participants will be administered 400 mg fluconazole followed by 200 mg fluconazole once daily from Days 12 to 26. During this time a single dose of 10 mg lemborexant will be administered following an overnight fast of at least 10 hours along with fluconazole on Day 15 only.
  Interventions: Drug: lemborexant; Drug: fluconazole

INTERVENTIONS:
Drug: lemborexant — oral tablet
  Other Names: E2006
Drug: Loestrin — oral tablet
  Arms: Part 1: Lemborexant plus Loestrin
Drug: famotidine — oral tablet
  Arms: Part 2: Lemborexant plus Famotidine
Drug: fluconazole — oral tablet
  Arms: Part 3: Lemborexant plus Fluconazole

SUMMARY:
This study will be conducted to evaluate the effect of lemborexant 10 milligrams (mg) (at steady state) on the pharmacokinetics (PK) of a single-dose combined oral contraceptive, Loestrin 1.5/30 (containing 0.030 mg of ethinyl estradiol and 1.5 mg of norethindrone), and to evaluate the effect of fluconazole 200 mg (at steady state) and a single dose of famotidine 40 mg (an H2 blocker) on the PK of a single oral dose of lemborexant 10 mg.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for All Participants (Part 1 - Oral Contraceptive; Part 2 - Famotidine; Part 3 - Fluconazole)

Participants who meet all of the following inclusion criteria will be eligible for participation in the study:

* Body mass index >18 and ≤32 kilograms per meters squared at Screening
* Are willing and able to comply with all aspects of the protocol
* Provide written informed consent

Additional Inclusion Criteria for Part 1 - Oral Contraceptive

* Healthy female participants, ages 18 to 44 years old (inclusive) at Screening
* Must not be taking any form of hormonal contraceptives, including hormonal intra-uterine device, for at least 8 weeks prior to dosing

Additional Inclusion Criteria (Part 2 - Famotidine; Part 3 - Fluconazole)

-Healthy male or female, age ≥18 years and ≤55 years old at the time of informed consent

Exclusion Criteria:

* Known contraindication to Loestrin (only for Part 1), to Famotidine (only for Part 2), or to Fluconazole (only for Part 3)
* Females who are breastfeeding or pregnant at Screening or Baseline.
* Females of childbearing potential. NOTE: All females will be considered to be of childbearing potential unless they are postmenopausal (amenorrheic for at least 12 consecutive months, in the appropriate age group, and without other known or suspected cause) or have been sterilized surgically (i.e., bilateral tubal ligation, total hysterectomy, or bilateral oophorectomy, all with surgery at least 1 month before dosing).
* Clinically significant illness that requires medical treatment within 8 weeks or a clinically significant infection that requires medical treatment within 4 weeks of dosing
* Presence of significant illness that requires treatment or may influence the study assessments (e.g. psychiatric disorders, disorders of the gastrointestinal tract, liver, kidney, respiratory system, endocrine system, hematological system, neurological system, cardiovascular system, or a congenital abnormality)
* Any history of abdominal surgery that may affect PK profiles of lemborexant (eg, hepatectomy, nephrectomy, digestive organ resection) at Screening
* Any other clinically abnormal symptom or organ impairment found by medical history, physical examinations, vital signs, electrocardiogram (ECG) finding, or laboratory test results that requires medical treatment at Screening or Baseline
* A prolonged QT/corrected QT (QTc) interval (QTc >450 milliseconds) demonstrated on ECG at Screening or Baseline
* Persistent systolic blood pressure (BP) >160 millimeters of mercury (mmHg) or diastolic BP >100 mmHg at Screening or Baseline (based on BP measured on at least 3 occasions over 2 weeks)
* Persistent heart rate (HR) of <50 beats per minute (beats/min) or >90 beats/min at Screening or Baseline (based on HR measured on at least 3 occasions over 2 weeks)
* Known history of clinically significant drug allergy at Screening or Baseline
* Known history of food allergies or presently experiencing significant seasonal or perennial allergy at Screening or Baseline
* Known to be human immunodeficiency virus positive
* Active viral hepatitis (B or C) as demonstrated by positive serology at Screening
* History of drug or alcohol dependency or abuse within the 2 years before Screening
* Participants who smoke or have used tobacco or nicotine-containing products within 4 weeks before dosing
* Any suicidal ideation with intent with or without a plan at Screening or within 6 months of Screening (ie, for Part 1 answering "Yes" to questions 4 or 5 on the Suicidal Ideation section of the Columbia-Suicide Severity Rating Scale) or any suicidal behavior in the past 10 years.
* Currently enrolled in another clinical trial or used any investigational drug or device within 30 days (or 5 half-lives, whichever is longer) preceding informed consent
* Engagement in strenuous exercise within 2 weeks before check-in (e.g., marathon runners, weight lifters)
* Intake of caffeinated beverages or caffeinated food within 72 hours before dosing and during the course of the study
* Intake of food supplements (including herbal preparations), foods, or beverages that may affect cytochrome P4503A4 enzyme (e.g., alcohol, grapefruit, grapefruit juice, grapefruit-containing beverages, apple or orange juice, vegetables from the mustard green family [e.g., kale, broccoli, watercress, collard greens, kohlrabi, Brussels sprouts, mustard], and charbroiled meats) within 1 week before dosing
* Intake of herbal preparations containing St. John's Wort within 4 weeks before dosing
* Intake of prescription or over-the-counter medications within 14 days (or 5 half-lives, whichever is longer) before dosing unless the Principal Investigator and medical monitor consider that they do not compromise participant safety or study assessments
* A positive urine drug test, a positive breathalyzer alcohol test, or, if appropriate, a positive serum pregnancy test

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2018-02-05 (Actual); Primary Completion 2018-03-23 (Actual); Study Completion 2018-03-23 (Actual)

PRIMARY OUTCOMES:
Part 1 (Lemborexant plus Loestrin): Mean maximum observed concentration (Cmax) of lemborexant and metabolites | Blood samples for lemborexant and metabolite assessment will be obtained at predose and 0.5 (30 minutes), 1, 1.5, 2, 3, 4, 5, 6, 8, 12, and 24 hours postdose on Days 14 and 15.
Part 1 (Lemborexant plus Loestrin): Mean predose drug concentration (Cmin) of lemborexant and metabolites | Blood samples for lemborexant and metabolite assessment will be obtained at predose and 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, and 24 hours postdose on Days 14 and 15.
Part 1 (Lemborexant plus Loestrin): Mean time to reach maximum (peak) drug concentration following drug administration (Tmax) of lemborexant and metabolites | Blood samples for lemborexant and metabolite assessment will be obtained at predose and 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, and 24 hours postdose on Days 14 and 15.
Part 1 (Lemborexant plus Loestrin): Mean area under the concentration-time curve from zero time to 24 hours postdose (AUC[0-24h]) of lemborexant and metabolites | Blood samples for lemborexant and metabolite assessment will be obtained at predose and 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, and 24 hours postdose on Days 14 and 15.
Part 2 (Lemborexant plus Famotidine): Mean Cmax of lemborexant and metabolites | Blood samples for lemborexant and metabolite assessment will be obtained at predose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72, 120, 168, and 216 hours after dosing on Days 1 and 15.
Part 2 (Lemborexant plus Famotidine): Mean Tmax of lemborexant and metabolites | Blood samples for lemborexant and metabolite assessment will be obtained at predose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72, 120, 168, and 216 hours after dosing on Days 1 and 15.
Part 2 (Lemborexant plus Famotidine): Mean AUC(0-24h) of lemborexant and metabolites | Blood samples for lemborexant and metabolite assessment will be obtained at predose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72, 120, 168, and 216 hours after dosing on Days 1 and 15.
Part 2 (Lemborexant plus Famotidine): Mean AUC from zero time to 72 hours postdose (AUC[0-72h]) of lemborexant and metabolites | Blood samples for lemborexant and metabolite assessment will be obtained at predose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72, 120, 168, and 216 hours after dosing on Days 1 and 15.
Part 2 (Lemborexant plus Famotidine): Mean AUC from zero time to last measurable time (AUC[0-t]) of lemborexant and metabolites | Blood samples for lemborexant and metabolite assessment will be obtained at predose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72, 120, 168, and 216 hours after dosing on Days 1 and 15.
Part 2 (Lemborexant plus Famotidine): Mean AUC from zero time extrapolated to infinite time (AUC[0-inf]) of lemborexant and metabolites | Blood samples for lemborexant and metabolite assessment will be obtained at predose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72, 120, 168, and 216 hours after dosing on Days 1 and 15.
Part 2 (Lemborexant plus Famotidine): Mean terminal elimination half-life (t1/2) of lemborexant and metabolites following the last dose | Blood samples for lemborexant and metabolite assessment will be obtained at predose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72, 120, 168, and 216 hours after dosing on Days 1 and 15.
Part 3 (Lemborexant plus Fluconazole): Mean Cmax of lemborexant and metabolites | Blood samples for lemborexant and metabolite assessment will be obtained on Days 1 to 27.
  Day 1 at predose and at approximately 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 12 hours postdose. At approximately 24, 48, and 72 (Days 2 to 4); 120 (Day 6); 168 (Day 8); 216 (Day 10) hours after the first dose. Day 15 at predose and at approximately 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 12 hours after the second dose. At approximately 24, 48, and 72 (Days 16 to 18); 120 (Day 20); 168 (Day 22); 216 (Day 24); 288 (Day 27) hours after the second dose.
Part 3 (Lemborexant plus Fluconazole): Mean Tmax of lemborexant and metabolites | Blood samples for lemborexant and metabolite assessment will be obtained on Days 1 to 27.
  Day 1 at predose and at approximately 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 12 hours postdose. At approximately 24, 48, and 72 (Days 2 to 4); 120 (Day 6); 168 (Day 8); 216 (Day 10) hours after the first dose. Day 15 at predose and at approximately 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 12 hours after the second dose. At approximately 24, 48, and 72 (Days 16 to 18); 120 (Day 20); 168 (Day 22); 216 (Day 24); 288 (Day 27) hours after the second dose.
Part 3 (Lemborexant plus Fluconazole): Mean AUC(0-24h) of lemborexant and metabolites | Blood samples for lemborexant and metabolite assessment will be obtained on Days 1 to 16.
  Day 1 at predose and at approximately 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 12 hours postdose. At approximately 24 (Day 2) hours after the first dose. Day 15 at predose and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 12 hours after the second dose. At approximately 24 (Day 16) hours after the second dose.
Part 3 (Lemborexant plus Fluconazole): Mean AUC(0-72h) of lemborexant and metabolites | Blood samples for lemborexant and metabolite assessment will be obtained on Days 1 to 18.
  Day 1 at predose and at approximately 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 12 hours postdose. At approximately 24, 48, and 72 (Days 2 to 4) hours after the first dose. Day 15 at predose and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 12 hours after the second dose. At approximately 24, 48, 72 hours (Days 16 to 18 after the second dose).
Part 3 (Lemborexant plus Fluconazole): Mean AUC(0-t) of lemborexant and metabolites | Blood samples for lemborexant and metabolite assessment will be obtained on Days 1 to 27.
  Day 1 at predose and at approximately 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 12 hours postdose. At approximately 24, 48, and 72 (Days 2 to 4); 120 (Day 6); 168 (Day 8); 216 (Day 10) hours after the first dose. Day 15 at predose and at approximately 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 12 hours after the second dose. At approximately 24, 48, and 72 (Days 16 to 18); 120 (Day 20); 168 (Day 22); 216 (Day 24); 288 (Day 27) hours after the second dose.
Part 3 (Lemborexant plus Fluconazole): Mean AUC(0-inf) of lemborexant and metabolites | Blood samples for lemborexant and metabolite assessment will be obtained on Days 1 to 27.
  Day 1 at predose and at approximately 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 12 hours postdose. At approximately 24, 48, and 72 (Days 2 to 4); 120 (Day 6); 168 (Day 8); 216 (Day 10) hours after the first dose. Day 15 at predose and at approximately 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 12 hours after the second dose. At approximately 24, 48, and 72 (Days 16 to 18); 120 (Day 20); 168 (Day 22); 216 (Day 24); 288 (Day 27) hours after the second dose.
Part 3 (Lemborexant plus Fluconazole): Mean t1/2 of lemborexant and metabolites following last dose | Blood samples for lemborexant and metabolite assessment will be obtained on Days 1 to 27.
  Day 1 at predose and at approximately 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 12 hours postdose. At approximately 24, 48, and 72 (Days 2 to 4); 120 (Day 6); 168 (Day 8); 216 (Day 10) hours after the first dose. Day 15 at predose and at approximately 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 12 hours after the second dose. At approximately 24, 48, and 72 (Days 16 to 18); 120 (Day 20); 168 (Day 22); 216 (Day 24); 288 (Day 27) hours after the second dose.

CONTACTS AND LOCATIONS:
Locations (1):
- Worldwide Clinical Trials, San Antonio, Texas, United States